CLINICAL TRIAL: NCT05477095
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, First-in-Human Study to Evaluate the Safety, Tolerability, and Immunogenicity of UBITh® CGRP Immunotherapy (UB-313) in Healthy Participants
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Immunogenicity of UB-313 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxxinity, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UB-313-101
Record Dates: First submitted 2022-07-20; First posted 2022-07-28 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- UB-313 Cohort 1 (Experimental): UB-313 100mcg administered by intramuscular (IM) injection at Week 0, Week 4 and Week 12
  Interventions: Biological: UB-313
- UB-313 Cohort 2 (Experimental): UB-313 300mcg administered by IM injection at Week 0 and 100mcg at Week 4 and Week 12
  Interventions: Biological: UB-313
- UB-313 Cohort 3 (Experimental): UB-313 300mcg administered by IM injection at Week 0, Week 4 and Week 12
  Interventions: Biological: UB-313
- UB-313 Cohort 4 (Experimental): UB-313 600mcg administered by IM injection at Week 0 and 100mcg at Week 4 and Week 12
  Interventions: Biological: UB-313
- Placebo Comparator (Placebo Comparator): Placebo (normal saline), administered by IM injection at Week 0, Week 4 and Week 12
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: UB-313 — A synthetic peptide-based immunotherapy
  Arms: UB-313 Cohort 1; UB-313 Cohort 2; UB-313 Cohort 3; UB-313 Cohort 4
Biological: Placebo — Normal saline
  Arms: Placebo Comparator

SUMMARY:
This first in-human (FIH) study of UB-313, an anti-calcitonin gene-related peptide based immunotherapeutic candidate, is designed to assess the safety, tolerability, and immunogenicity of 4 selected UB-313 dose regimens in healthy adults.

DETAILED DESCRIPTION:
This is a single-site, randomized, double-blind, placebo-controlled, multidose regimen, FIH study of UB-313, an anti-CGRP peptide-based immunotherapy candidate. The double-blind period will include dose escalation and cohort staggering for up to 4 planned dose levels of UB-313 or placebo in 4 cohorts of healthy participants. All eligible participants will be enrolled in the study for up to 44 weeks, consisting of IM injections of UB-313 or placebo at Week 0 (Baseline, Day 1), Week 4, and Week 12. The End of Treatment (EoT) is defined as Week 16, followed by a follow-up period up to Week 44.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female aged 18 to 55 years old, inclusive, at time of informed consent.
* Has a body mass index between 18 and 30 kg/m2, inclusive at Screening, and with a minimum weight of 50 kg.
* Male participants and their partners of childbearing potential must commit to the use of highly effective contraceptives for the study duration and for at least 12 weeks after the last dose. Men must refrain from donating sperm during this same period.
* Female participants must be of nonchildbearing potential, or, for women of childbearing potential, must be willing to practice highly effective contraception throughout the duration of the study and for at least 24 weeks following the last dose.
* Other inclusion criteria apply

Exclusion Criteria:

* Has a history of clinically significant medical or psychiatric conditions, which in the opinion of the Investigator may compromise the participant's safety or the scientific value of the study, posing an unacceptable risk to the participant or interfere with the participant's ability to comply with study procedures or abide by study restrictions.
* Presents any concern by the Investigator regarding safe participation in the study or for any other reason (including contraindication to MRI) that the Investigator considers the participant inappropriate for participation in the study.
* Has a recent history (within the past year of Screening) of migraine headache.
* Has unsuitable skin characteristics for the dermal capsaicin challenge as determined by the Investigator.
* Has not demonstrated at least a 100% increase in dermal blood flow following capsaicin challenge as part of Screening procedures and measured through laser speckle contrast imaging.
* Other exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Vaxxinity, Inc.
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UB-313 Cohort 1 | UB-313 Cohort 2 | UB-313 Cohort 3 | UB-313 Cohort 4 | Placebo Comparator
Started | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 8
Not Completed | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UB-313 Cohort 1 | UB-313 Cohort 2 | UB-313 Cohort 3 | UB-313 Cohort 4 | Placebo Comparator | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (13.66) | 32.5 (8.52) | 31.6 (11.92) | 30.4 (7.87) | 26.0 (8.88) | 31.1 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 5 | 4 | 21
  Male | 5 | 5 | 2 | 3 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 8 | 8 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.39 (3.388) | 23.58 (1.834) | 24.29 (3.624) | 21.88 (2.384) | 23.68 (2.600) | 23.76 (2.931)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: The number and percentage of participants with TEAEs were tabulated.
Time Frame: 44 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | UB-313 Cohort 1 | UB-313 Cohort 2 | UB-313 Cohort 3 | UB-313 Cohort 4 | Placebo Comparator
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants | 7 | 8 | 6 | 8 | 7

2. Primary Outcome: Immunogenicity Measured by Serum Anti-CGRP Antibodies.
Description: Immunogenicity measured by blood anti-CGRP antibody titers, reported as Optical Density (OD) of 1:25 dilution.
Time Frame: Weeks 0, 1, 4, 5, 8, 12, 13, 16, 20, 28, 36 and 44; Week 0, Week 16 and Week 44 are reported
Measure: Mean (Standard Deviation); unit: Optical Density (OD)
Arm/Group | UB-313 Cohort 1 | UB-313 Cohort 2 | UB-313 Cohort 3 | UB-313 Cohort 4 | Placebo Comparator
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8
Optical Density (OD)
  Week 0 (Baseline) | 0.5161 (0.1697) | 0.4720 (0.1688) | 0.6024 (0.2292) | 0.5495 (0.0994) | 0.4900 (0.0862)
  Week 16 (EoT) | 2.7271 (1.2042) | 2.1900 (1.0378) | 3.2903 (0.7628) | 3.0731 (0.9075) | 0.4776 (0.0861)
  Week 44 (EoS) | 1.4449 (0.8055) | 1.2225 (0.5760) | 1.7653 (0.9176) | 1.5401 (0.7779) | 0.5614 (0.1321)

3. Secondary Outcome: Pharmacodynamics of the Immune Response Measured by Capsaicin-induced Increase in Dermal Blood Flow
Description: Number of Participants with inhibition of capsaicin-induced increase in dermal blood flow
Time Frame: Weeks 0, 4, 8, 12, 16, 20
Measure: Count of Participants; unit: Participants
Arm/Group | UB-313 Cohort 1 | UB-313 Cohort 2 | UB-313 Cohort 3 | UB-313 Cohort 4 | Placebo Comparator
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8
Participants
  Baseline | 0 | 1 | 0 | 0 | 0
  Week 4 | 1 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0
  Week 12 | 0 | 0 | 0 | 0 | 1
  Week 16 | 0 | 0 | 0 | 0 | 1
  Week 20 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the length of the participants enrollment in the study which was 44 weeks.
Description: Definition does not differ.
Arm/Group | UB-313 Cohort 1 | UB-313 Cohort 2 | UB-313 Cohort 3 | UB-313 Cohort 4 | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8 | 6/8 | 8/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UB-313 Cohort 1 (N=8) | UB-313 Cohort 2 (N=8) | UB-313 Cohort 3 (N=8) | UB-313 Cohort 4 (N=8) | Placebo Comparator (N=8)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 | 1 | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 2
General disorders and administration site conditions (General disorders) | 4 | 5 | 5 | 7 | 2
Injection site pain (General disorders) | 3 | 4 | 2 | 7 | 1
Fatigue (General disorders) | 4 | 2 | 2 | 3 | 1
Infections and infestations (Infections and infestations) | 4 | 4 | 6 | 5 | 5
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 | 2 | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 4 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 1
Nervous system disorders (Nervous system disorders) | 5 | 4 | 4 | 6 | 5
Headache (Nervous system disorders) | 5 | 4 | 4 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT05477095/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT05477095/SAP_001.pdf